CLINICAL TRIAL: NCT07368608
Title: A Randomized, Double-blind, Placebo-controlled Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Subcutaneous BEBT-701 in Patients With Mild to Moderate Hypertension and Elevated LDL-C
Brief Title: A Study of BEBT-701 in Patients With Mild to Moderate Hypertension and Elevated Low-Density Lipoprotein Cholesterol（LDL-C）
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBMT-701-P01
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mild to Moderate Hypertension and Elevated Low-Density Lipoprotein Cholesterol
Keywords: BEBT-701; Safety; Tolerability; Pharmacokinetics; Preliminary Efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I Single-Dose Cohorts (BEBT-701) (Experimental): Phase I: Five predefined dose cohorts are planned. In each cohort, the first two subjects (randomized 1:1 to active drug or placebo) are dosed in a sentinel fashion. Only after these two subjects have completed at least 48 h of safety observation and the investigator has confirmed acceptable tolerability will the remaining six subjects be enrolled and dosed at a 5:1 ratio (active drug : placebo). Enrollment and dosing of the next higher dose cohort will begin only after every subject in the preceding cohort has completed a minimum 2-week safety observation period and the safety data are judged acceptable.
  Interventions: Drug: BEBT-701 Injection
- Phase I Single-Dose Cohorts (Placebo) (Placebo Comparator): Phase I: Five predefined dose cohorts are planned. In each cohort, the first two subjects (randomized 1:1 to active drug or placebo) are dosed in a sentinel fashion. Only after these two subjects have completed at least 48 h of safety observation and the investigator has confirmed acceptable tolerability will the remaining six subjects be enrolled and dosed at a 5:1 ratio (active drug : placebo). Enrollment and dosing of the next higher dose cohort will begin only after every subject in the preceding cohort has completed a minimum 2-week safety observation period and the safety data are judged acceptable.
  Interventions: Drug: BEBT-701 Injection Placebo（0.9% Sodium Chloride Injection）
- Phase II Multiple-Dose Cohorts (BEBT-701) (Experimental): Phase II: Based on the preliminary safety, PK, and PD data from the Phase I single-dose study, three dose levels will be selected for further evaluation. Eligible subjects will be randomized in a 1:1:1:1 ratio to one of the three pre-specified active doses or to placebo.
  Interventions: Drug: BEBT-701 Injection
- Phase II Multiple-Dose Cohorts (Placebo) (Placebo Comparator): Phase II: Based on the preliminary safety, PK, and PD data from the Phase I single-dose study, three dose levels will be selected for further evaluation. Eligible subjects will be randomized in a 1:1:1:1 ratio to one of the three pre-specified active doses or to placebo.
  Interventions: Drug: BEBT-701 Injection Placebo（0.9% Sodium Chloride Injection）

INTERVENTIONS:
Drug: BEBT-701 Injection — Phase I: The starting dose of BEBT-701 injection is 100 mg; the single subcutaneous doses are 100 mg, 200 mg, 400 mg, 800 mg, and 1200 mg.
  Phase II: Based on the preliminary Phase I findings, three dose levels will be selected for the Phase II study, with BEBT-701 injection administered subcutaneously on Day 1 and Day 85.
  Arms: Phase I Single-Dose Cohorts (BEBT-701); Phase II Multiple-Dose Cohorts (BEBT-701)
Drug: BEBT-701 Injection Placebo（0.9% Sodium Chloride Injection） — Phase I：BEBT-701 injection placebo, administered as a single subcutaneous dose. Phase II:BEBT-701 injection placebo administered subcutaneously on Day 1 and Day 85.
  Arms: Phase I Single-Dose Cohorts (Placebo); Phase II Multiple-Dose Cohorts (Placebo)

SUMMARY:
This Phase I/II clinical trial is designed to evaluate, through a single-dose Phase I segment and a multiple-dose Phase II segment, the safety/tolerability, pharmacokinetic (PK) profile, and pharmacodynamic (PD) characteristics of BEBT-701 administered by subcutaneous injection in patients with mild to moderate hypertension and elevated LDL-C , and to explore its preliminary efficacy.

DETAILED DESCRIPTION:
This study employs an integrated Phase I/II seamless adaptive design. Stage 1 is a single-dose Phase I component, randomized, double-blind, and placebo-controlled, with five pre-specified dose cohorts starting at 100 mg. Its primary objectives are to characterize the safety, tolerability, PK, PD, and preliminary efficacy of single-dose BEBT-701 across the planned dose range, thereby providing critical input for dose and dosing-interval selection for Stage 2.

After a 2- to 4-week observation period following the last Phase I cohort, three doses (preliminary) will be selected from the accumulated data to initiate Stage 2, a multiple-dose Phase II segment. This stage is a randomized, double-blind, parallel-group comparison of three active dose levels versus placebo. Placebo recipients will crossover to active treatment at Week 12 after the second dose; active-arm subjects will enter a double-blind extension after completing the 24-week post-second-dose visit, enabling collection of longer-term safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 60 years (inclusive).
2. Subjects with essential hypertension who are either treatment-naive or have remained off any antihypertensive medication for ≥ 30 days prior to screening and in whom the investigator deems no additional antihypertensive therapy necessary during the study period.
3. Body-mass index (BMI) 18.6-30kg/m² (inclusive); body weight ≥ 50 kg for men and ≥ 45 kg for women.
4. Has maintained a stable diet for at least 4 weeks before screening and has no plan to make a clinically significant change in diet or body weight during the study (a change > 10 % is considered significant).
5. Agrees to use a highly effective method of contraception and to avoid becoming a parent from enrollment until 12 months after the last dose.
6. Able to understand the study requirements, willing to comply, and provides written informed consent.

   Phase I subjects must simultaneously meet the following criteria:
7. At screening and within 24 h before randomization, the 24-h ambulatory blood-pressure monitoring shows mean systolic blood pressure (SBP) > 130 mmHg and < 150 mmHg.
8. At screening and baseline, fasting serum LDL-C is ≥ 100 mg/dL (2.6 mmol/L) and < 190 mg/dL (4.9 mmol/L) in subjects who are either lipid-lowering-therapy-naive or have not received any lipid-lowering drug within 30 days before screening and whom the investigator judges will not require any additional lipid-lowering therapy during the study.

   Phase II subjects must simultaneously meet the following criteria:
9. At screening and within 24h before randomization, 24-h ambulatory blood-pressure monitoring must show mean SBP > 130 mmHg and < 160 mmHg.
10. At screening and baseline, fasting serum LDL-C ≥ 100 mg/dL (2.6 mmol/L). Subjects already on statin therapy must have been on a stable statin dose and regimen for at least 30 days prior to screening and must have no planned changes to their statin treatment during the study.

Exclusion Criteria:

1. Any history of severe illness-apart from hypertension and hyperlipidemia-that in the investigator's opinion could influence trial outcomes, including but not limited to diseases of the circulatory system (e.g., orthostatic hypotension, NYHA class II-IV heart failure, aortic stenosis, major aortic aneurysm or dissection, hypertensive encephalopathy, acute stroke, transient ischemic attack, acute myocardial infarction, significant arrhythmias), endocrine, neurologic, gastrointestinal, genitourinary, hematologic, immunologic, psychiatric, or metabolic disorders.
2. History of allergic disease or atopic diathesis (≥3 drug or food allergies), or known hypersensitivity to oligonucleotide-based therapeutics.
3. Use of anti-PCSK9 or anti-AGT antibody agents within 6 months before screening, or of PCSK9- or AGT-targeted oligonucleotide drugs within 12 months before screening.
4. Malignancy within 5 years before informed-consent signature (exceptions: adequately resected and cured basal- or squamous-cell skin carcinoma, cervical carcinoma in situ, or other cancers considered cured by surgery alone).
5. Left-ventricular ejection fraction (LVEF) < 40% at screening; or significant aortic or peripheral vascular disease, or any vascular condition requiring surgical intervention.
6. Type 1 diabetes, or type 2 diabetes with inadequate glycaemic control (HbA1c ≥ 8%).
7. Major surgery within 6 months before dosing, or planned major surgery during the study period.
8. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² (by simplified MDRD equation) or urine albumin-to-creatinine ratio (UACR) > 300 mg/g at screening.
9. At screening, any of the following laboratory abnormalities: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin(TBIL),gamma-glutamyl transferase(GGT), or alkaline phosphatase(ALP) > 1.5 × upper limit of normal (ULN), or serum potassium > 5.5 mmol/L (one repeat measurement permitted).
10. Mean 24-h ambulatory diastolic blood pressure (DBP) > 110 mmHg at screening and/or within 24 h prior to randomization (one repeat measurement permitted).
11. QT/QTc prolongation at screening or baseline: QT interval corrected by Fridericia's formula (QTcF)≥ 450 ms (men) or ≥ 460 ms (women).
12. Positive serology for HBsAg, anti-hepatitis C virus(HCV), HCV core antigen, anti-human immunodeficiency virus (HIV), or Treponema pallidum antibody; if Treponema pallidum antibody is positive, a confirmatory rapid plasma reagin(RPR) test is required and must also be positive.
13. Known or suspected secondary hypertension, including but not limited to bilateral renal-artery stenosis, primary aldosteronism, pheochromocytoma, polycystic kidney disease, or drug-induced hypertension.
14. Occupations involving hazardous operations such as piloting vessels or working at height.
15. Subcutaneous-injection intolerance, or prominent abdominal scarring, tattoos, or other conditions that could materially interfere with study-drug administration or the assessment of local tolerability.
16. Blood loss or donation > 400 mL within 3 months before dosing (menstrual bleeding excluded) and/or platelet donation within 2 weeks.
17. Use, within 28 days before dosing, of any drug, nutraceutical, vitamin, or dietary supplement known to affect lipid metabolism.
18. History of drug abuse or positive urine drug screen, and/or use of illicit drugs within 3 months before screening, and/or habitual use of any psychoactive substance (including herbal preparations).
19. Average daily consumption > 5 cigarettes (or equivalent e-cigarette use) within 3 months before screening and/or unwillingness to abstain from all tobacco products during the study.
20. Regular alcohol consumption within 6 months before screening (i.e., > 14 units/week; 1 unit = 360 mL of 5% beer, 45 mL of 40% spirits, or 150 mL of 12% wine) and inability to comply with alcohol-restriction requirements during the study.
21. Daily intake of excessive tea, coffee, and/or caffeine-containing beverages (≥ 8 cups/day; 1 cup = 250 mL) within 1 month before screening.
22. Participation in any clinical trial within 3 months before screening (12 months for oligonucleotide investigational drugs).
23. Subjects who, for any other reason, are unlikely to complete the study or whom the investigator deems should not be enrolled.
24. Pregnant or lactating women.
25. History of syncope within 3 months before screening.
26. Receipt of a live vaccine within 4 weeks before screening or planned live-vaccine administration during the study.
27. Use of long-acting estrogen and/or progestin injections or implants within 6 months before dosing.
28. Women of child-bearing potential who engaged in unprotected intercourse with a partner within 28 days before dosing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events (AEs) | Up to 36 months
  Occurrence of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V5.0).
Low-Density Lipoprotein Cholesterol(LDL-C) | Up to 24 weeks
  Percentage change from baseline in LDL-C after dosing.
24hour-Ambulatory Blood Pressure Monitoring（24h-ABPM） | Up to 24weeks
  Change from baseline in mean 24h-ABPM systolic blood pressure (SBP) after dosing.

SECONDARY OUTCOMES:
AUC0-∞ | Phase I:From pre-dose to 72 h post-dose on Day 1; Phase II:From pre-dose to 72 h post-dose on Day 1and Day 85.
  The area under the plasma concentration-time curve from time zero to infinity.
Cmax | Phase I:From pre-dose to 72 h post-dose on Day 1; Phase II:From pre-dose to 72 h post-dose on Day 1and Day 85.
  The maximum plasma drug concentration
Tmax | Phase I:From pre-dose to 72 h post-dose on Day 1; Phase II:From pre-dose to 72 h post-dose on Day 1and Day 85.
  The time to reach maximum plasma drug concentration
t1/2 | Phase I:From pre-dose to 72 h post-dose on Day 1; Phase II:From pre-dose to 72 h post-dose on Day 1and Day 85.
  The time for plasma drug concentration to halve
Blood pressure-related parameters | Up to 24 weeks
  Percentage change from baseline in mean 24-h ABPM SBP; Change from baseline in mean 24-h ABPM SBP; Change from baseline and percentage change from baseline in mean 24-h ABPM DBP,standard daytime mean SBP and DBP (6 a.m.-10 p.m.), standard nighttime mean SBP and DBP (10 p.m.-6 a.m.)； Change from baseline and percentage change from baseline in office seated SBP, DBP, and mean arterial pressure (MAP).
Lipid-related parameters | Up to 24 weeks
  Percentage change from baseline in LDL-C；Change from baseline and percentage change from baseline in total cholesterol (TC), high-density-lipoprotein cholesterol (HDL-C), non-high-density-lipoprotein cholesterol (non-HDL-C), very-low-density-lipoprotein cholesterol (VLDL-C), apolipoprotein B, apolipoprotein A1, triglycerides, and lipoprotein(a).
Angiotensinogen(AGT) | Up to 36 weeks
  Change from baseline and percentage change from baseline in AGT.
Proprotein convertase subtilisin/kexin type 9 (PCSK9) | Up to 36 weeks
  Change from baseline and percentage change from baseline in PCSK9.

OTHER OUTCOMES:
Immunogenicity parameters | Up to 36 weeks
  Anti-drug antibodies(ADA), interleukin-2(IL-2), interleukin-4(IL-4), interleukin-6(IL-6), interleukin-10(IL-10), interferon-gamma(IFN-γ), tumor necrosis factor-alpha(TNF-α), complement 3(C3)and complement 4(C4).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yuan, Ph.D, Principal Investigator — The Third Xiangya Hospital of Central South University; Guoping Yang, Ph.D, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China